CLINICAL TRIAL: NCT06961266
Title: A Phase 1b, Randomized, Double-blind, Sponsor-Unblinded, Placebo-Controlled 4-Way Crossover Study to Evaluate Efficacy, Safety, Tolerability, and Pharmacokinetics of JZP441 in Participants With Narcolepsy Type 1
Brief Title: A Study to Investigate Efficacy, Safety, Tolerability, and Pharmacokinetics of JZP441 Compared With Placebo in Participants With Narcolepsy Type 1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Jazz Pharmaceuticals Ireland Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: JZP441-105
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Narcolepsy
Keywords: Narcolepsy Type 1; JZP441
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled crossover study
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- JZP441 Dose Level 1 (Experimental): Participants with narcolepsy type 1 who are randomized to receive JZP441.
  Interventions: Drug: JZP441
- JZP441 Dose Level 2 (Experimental): Participants with narcolepsy type 1 who are randomized to receive JZP441.
  Interventions: Drug: JZP441
- JZP441 Dose Level 3 (Experimental): Participants with narcolepsy type 1 who are randomized to receive JZP441.
  Interventions: Drug: JZP441
- Placebo (Placebo Comparator): Participants with narcolepsy type 1 who are randomized to receive matching placebo.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: JZP441 — Administered orally
  Arms: JZP441 Dose Level 1; JZP441 Dose Level 2; JZP441 Dose Level 3
Drug: Matching Placebo — Administered orally
  Arms: Placebo

SUMMARY:
Narcolepsy is a sleep disorder in which patients are not able to maintain wakefulness or require treatment to maintain wakefulness during the daytime. Narcolepsy is a lifelong neurologic disease for which no cure has been clinically available. JZP441 is currently being developed for the treatment of narcolepsy type 1 (NT1). This study will assess the safety of efficacy of JZP441 in adult patients with NT1.

DETAILED DESCRIPTION:
This Phase 1b, randomized, double-blind, sponsor-unblinded, placebo-controlled 4-way crossover study will evaluate the efficacy, safety, tolerability, and pharmacokinetics (PK) of a range of JZP441 doses in participants with NT1. Changes in daytime sleepiness will be assessed via objective (MWT) and subjective (KSS, VAS for sleepiness) efficacy measures.

ELIGIBILITY:
Participants are eligible to be included in the study only if all of the following criteria apply:

1. Is 18 to 64 years of age inclusive at the time of signing the informed consent.
2. Has a physician diagnosis of NT1 according to ICSD-3-TR criteria
3. Has an average sleep latency of less than 15 minutes, as documented by the mean of the first 4 trials of the Baseline MWT, as determined by central assessment.
4. Has a minimum body weight of 50 kg for men and 45 kg for women and a BMI within the range 18.0 to 35.0 kg/m^2 (inclusive).
5. Participant agrees to the following based on sex assigned at birth.

   1. Male participants are eligible to participate if they agree to the following during the study intervention period and for at least 90 days after the last dose of study intervention:

      * Refrain from donating sperm
      * Use contraception /barrier as specified in the protocol
   2. Female participants are eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

      * Is a woman of non-childbearing potential (WONCBP) OR
      * Is a WOCBP and using a contraceptive method that is highly effective during the study intervention period and until completion of the Safety Follow-up Period.
      * Male partners of WOCBP are required to use barrier protection, (eg, condoms) during the study intervention period and over the 90-day period after the last dose of study intervention.

        • A WOCBP must have a negative highly sensitive pregnancy test at screening and at check-in on Day -1 of each Treatment Visit, before the first dose of study intervention is administered.
      * If a urine test cannot be confirmed as negative, a serum pregnancy test is required.
6. Is capable of giving signed informed consent

Participants are excluded from the study if any of the following criteria apply:

1. Any other clinically relevant medical, behavioral, or psychiatric disorder other than NT1 that is associated with EDS.
2. History or presence of gastrointestinal (including gastric bypass surgery within the past 10 years), hepatic disease, untreated thyroid disease, or any other condition that may interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Presence of severe renal impairment, end-stage renal disease or BSA-adjusted calculated eGFR <60 mL/min.
4. Presence of cardiodynamic abnormalities defined as triplicate 12-lead ECG
5. History or evidence of any of the following: myocardial infarction, cardiac surgery revascularization, unstable angina, cerebrovascular accident or stroke or TIA, pacemaker, atrial fibrillation, flutter, syncope in the past 2 years from a cardiac etiology or unexplained syncope or non-sustained or sustained VT. Angina pectoris greater than Class 1, CHF greater than NYHA Class 1, personal or family history of the Long QT Syndrome, Brugada syndrome, Wolff-Parkinson-White syndrome, any history of heart block, family history of sudden death.
6. Structural or functional heart abnormalities as determined by an echocardiogram performed within 6 months prior to screening, including LVEF <45%; moderate or greater aortic or mitral stenosis or regurgitation.
7. Presence or history of uncontrolled hypertension, systolic BP of at least 140 mmHg or diastolic BP of at least 90 mmHg (at Screening Visit, Baseline Visit, or prior to randomization).
8. Laboratory values (chemistry, hematology, and urinalysis) outside the laboratory reference range considered to be clinically significant by the investigator.
9. History of suicide attempt, current suicidal risk as determined from history, or presence of active suicidal ideation as indicated by a positive response to item 4 or item 5 on the C-SSRS (within the past 6 months).
10. Current major depressive episode or presence of uncontrolled anxiety disorder according to DSM-5 criteria. Participants with stable treated depression and/or anxiety are allowed.
11. Current or history of psychotic or bipolar disorders, or any first degree relative with a history of schizophrenia-spectrum disorder or bipolar I disorder.
12. History (within the past year at screening) or presence of substance use disorder or alcohol use disorder per DSM-5 definition, known drug dependence, or seeking treatment for alcohol or substance use related disorder.
13. History of seizure disorder or a physical condition that would increase seizure risk.
14. History of ischemic event or a condition that elevates the participant's risk for an ischemic event
15. Evidence of untreated or inadequately treated sleep-disordered breathing
16. Concomitant or recent (within 5 half-lives) use of drugs that affect QT or QRS intervals, including sodium channel blockers.
17. Use of any medications that could affect the evaluation of EDS within a time period prior to the Baseline Visit corresponding to at least 5 half-lives of the drug(s) or planned use during the study.
18. Concomitant use of XYWAV, high sodium oxybate, or pitolisant. Other medications used for treatment of cataplexy (eg, antidepressants) are allowed.
19. Participation in another clinical study of an investigational drug (other than JZP441) or medical device within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention and throughout the duration of the study.
20. Habitual bedtime later than 1:00 AM over the last 6 months, per self-report.
21. Occupation requiring nighttime shift work or variable shift work.
22. Travel across 3 or more time zones within 1 week of Baseline Visit or planned through duration of treatment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Mean sleep latency of the first 4 sessions of the Maintenance of Wakefulness Test | 1, 3, 5, and 7 hours after the first dose of study intervention
  The MWT is the standard objective measure of an individual's ability to remain awake during the daytime in a darkened quiet environment and is commonly used to assess response to treatment. The MWT will be used to compare the pharmacodynamic response of JZP441 versus placebo. Sleep latency will be reported in minutes.

SECONDARY OUTCOMES:
Number of Participants Reporting Treatment-emergent Adverse Events | Baseline up to Week 11
  A treatment-emergent adverse event (TEAE) is defined as an adverse event (AE) that started, or worsened in severity or seriousness, following a dose of study intervention.
Pharmacokinetic Parameter Maximum Plasma Concentration | Day 1 (predose), 2, 4, 6, 8, 10, and 12 hours post first dose; Day 2 (24 hours) post first dose.
Pharmacokinetic Parameter Time to Maximum Plasma Concentration | Day 1 (predose), 2, 4, 6, 8, 10, and 12 hours post first dose; Day 2 (24 hours) post first dose.
Pharmacokinetic Parameter Area Under the Plasma Concentration Curve | Day 1 (predose), 2, 4, 6, 8, 10, and 12 hours post first dose; Day 2 (24 hours) post first dose.
Mean Score of the First 4 assessments of Karolinska Sleepiness Scale | 1, 3, 5, 7, 9 and 11 hours after first dose
  The Karolinska Sleepiness Scale (KSS) is a single-item, 9-point, self-administered questionnaire that measures a participant's subjective level of sleepiness (from "extremely alert" to "extremely sleepy, can't keep awake"). Scores generally decrease with longer periods of wakefulness, indicating that lower scores correlate with better outcomes.
Mean VAS Score For Sleepiness | 1, 3, 5, 7, 9 and 11 hours after first dose
  The self-reported VAS measure of sleepiness in the current study will be a retrospective measure of how sleepy the participant felt throughout the day, with anchors at each end of the line labeled as "0=not at all sleepy" to "100=very sleepy." Higher VAS scores indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Lead, Study Director — Jazz Pharmaceuticals
Locations (4):
- United States (4):
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Cincinnati, Ohio
  - Clinical Trial Site, Columbia, South Carolina
  - Clinical Trial Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
In accordance with ICMJE requirements, Jazz Pharmaceuticals may provide qualified external researchers access to individual participant data (IPD) and clinical trial data that underlie the results of this trial upon request. Qualified researchers can submit a request on https://www.jazzpharma.com/science/clinical-trial-data-sharing/ as outlined. Jazz Pharmaceuticals reserves the right not to consider a request. For inquiries about Jazz's data sharing policy contact clinicaldatasharing@jazzpharma.com.